CLINICAL TRIAL: NCT00927251
Title: Model 4296 Left Ventricular Lead Study
Brief Title: Model 4296 Left Ventricular (LV) Lead Study
Acronym: 4296
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4296
Record Dates: First submitted 2009-06-23; First posted 2009-06-24 (Estimated); Results first posted 2010-12-29 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2019-01

CONDITIONS: Heart Failure
Keywords: heart failure; cardiac pacing; cardiac resynchronization therapy; left ventricular lead
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Model 4296 LV Lead (Experimental): Non-randomized study
  Interventions: Device: Pacing Lead (Model 4296 LV Lead)

INTERVENTIONS:
Device: Pacing Lead (Model 4296 LV Lead) — Implant and follow-up of study device

SUMMARY:
This study is designed to show that a new lead, which paces the left bottom chamber (left ventricle) of the heart, is safe. Using a lead on the left side of the heart has been shown to potentially improve heart failure symptoms. The shape and size of this new lead may make it a good choice for patients or physicians.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, non-randomized design trial. All consented patients who meet all inclusion and no exclusion criteria may receive the investigational lead. The study design has statistical power to show safety at one-month after implant.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac Resynchronization Therapy (CRT)/Cardiac Resynchronization Therapy-Defibrillator (CRT-D) indications according to the European Society of Cardiology/American College of Cardiology/American Heart Association (ESC/ACC/AHA) guidelines
* On optimal medical treatment according to investigator opinion
* Indicated for implantable cardioverter defibrillator (ICD) if CRT-D is implanted
* Patient consent
* Geographically stable

Exclusion Criteria:

* Left Ventricular (LV) lead implant attempt in last 30 days
* Unstable angina or acute myocardial infarction (MI) in past 30 days
* Coronary artery bypass graft (CABG) or percutaneous transluminal coronary angioplasty (PTCA) in past 90 days
* Contraindicated for transvenous pacing
* Heart transplant
* Contraindicated for less than 1 milligram (mg) dexamethasone acetate
* Enrolled or intends to participate in concurrent drug and/or device study which would confound results
* Life expectancy shorter than duration of the study
* Exclusion criteria required by local law
* Unable to tolerate urgent thoracotomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Biffi, M.D., Principal Investigator — Policlinico S. Orsola-Malpighi in Bologna, Italy
Locations (16):
- Austria (2):
  - Linz
  - Vienna
- Oulu, Finland
- Germany (5):
  - Bad Rothenfelde
  - Essen
  - Heidelberg
  - Lüdenscheid
  - Ulm
- Delhi, India
- Italy (3):
  - Bologna
  - Pesaro
  - Rovigo
- Netherlands (2):
  - Breda
  - Eindhoven
- Bergen, Norway
- Košice, Slovakia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial began with the first subject enrollment on July 1, 2009 and subsequent first implant of the Model 4296 LV lead on July 2, 2009. A total of 90 subjects were enrolled in the study of which 82 were successfully implanted with a Model 4296 LV lead. Last enrollment took place on December 16, 2009.
Groups:
- Model 4296 LV Lead Study: This study is a prospective, multi-center, non-randomized, one-arm clinical trial using Objective Performance Criteria (OPC) to evaluate the safety and efficacy of the Model 4296 LV lead. The OPC based trial design is consistent with the designs used to evaluate all current market released Medtronic left ventricular leads. The Model 4296 LV lead is designed to provide physicians with acceptable unipolar pacing from two selectable electrodes.All subjects are planned to undergo a CRT system implant and will be followed through at least pre-hospital discharge and one month visit.
Period: Overall Study
Arm/Group | Model 4296 LV Lead Study
Started | 90
Completed | 82
Not Completed | 8
Not completed — Patients not implanted with 4296 lead | 8

BASELINE CHARACTERISTICS:
Arm/Group | Model 4296 LV Lead Study
Number analyzed (Participants) | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 69
Region of Enrollment [Number; unit: participants]
  Slovakia | 10
  Austria | 11
  Norway | 3
  Netherlands | 14
  Germany | 43
  Italy | 9
New York Heart Association Functional Classification [Number; unit: participants] — Class I No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, or dyspnea.
  Class II Slight limitation of physical activity. Comfortable at rest, but ordinary physical activity results in fatigue, palpitation, or dyspnea.
  Class III Marked limitation of physical activity. Comfortable at rest, but less than ordinary activity causes fatigue, palpitation, or dyspnea.
  Class IV Unable to carry out any physical activity without discomfort. Symptoms of cardiac insufficiency at rest. If any physical activity is undertaken, discomfort is increased.
  participants
    NYHA Class II | 3
    NYHA Class III | 86
    NYHA Class IV | 1
Left Ventricular Ejection Fraction [Mean (Standard Deviation); unit: Percentage (%)] — The Left Ventricular Ejection fraction is the percentage of blood ejected from the left ventricle with each heart beat.
  Percentage (%) | 25.6 (6.5)
QRS Duration [Mean (Standard Deviation); unit: milliseconds] | 159.0 (21.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Left Ventricular (LV)Lead Related Complications
Description: A LV lead related complication occurs when an invasive procedure is needed to correct an adverse event related to the LV lead.
Time Frame: Implant to one-month post implant
Population: All subjects implanted with the lead who had completed their one-month post-implant/or a later follow-up visit, or have had a complication by the one-month post-implant visit, were included in the analysis. A complication is defined as an Adverse Event that results in death, any termination of significant device function or invasive intervention
Measure: Number; unit: participants
Arm/Group | Model 4296 LV Lead Study
Number analyzed (Participants) | 67
participants | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the total duration of the study (from patient signing informed consent until study exit/study closure).The data provided shows adverse events reported until the last enrolled patient had completed his/her one month visit.
Description: At each follow up, patients were asked whether an adverse event had occurred.A patient was not allowed to exit the study until all relevant implant related AEs were resolved or determined to be irresolvable.
Arm/Group | Model 4296 LV Lead Study
Serious Adverse Events (participants affected / at risk) | 16/90
Other Adverse Events (participants affected / at risk) | 26/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Model 4296 LV Lead Study (N=90)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Catheter infection (Infections and infestations) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Decompensated heart failure (Cardiac disorders) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1)
Exit block (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture subtrochanteric (Injury, poisoning and procedural complications) | 1 (1)
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Lead dislodgement (Injury, poisoning and procedural complications) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuropneumonia (Infections and infestations) | 1 (1)
Syncope vasovagal (Nervous system disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 2 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Model 4296 LV Lead Study (N=90)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 3 (3)
Conjunctivitis (Eye disorders) | 1 (1)
Device lead issue (Injury, poisoning and procedural complications) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Drug side effect (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Gynecomastia (Reproductive system and breast disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Inappropriate phrenic nerve stimulation (Injury, poisoning and procedural complications) | 10 (12)
Inappropriate stimulation of diaphragm (Injury, poisoning and procedural complications) | 1 (1)
Infection urinary tract (Infections and infestations) | 1 (1)
Lead dislodgement (Injury, poisoning and procedural complications) | 1 (1)
Loss of sensation (Nervous system disorders) | 1 (1)
Medical device pain (Injury, poisoning and procedural complications) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Recurrent atrial fibrillation (Cardiac disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Tachyarrhtythmia absoluta (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, contracts allow investigators to publish study results per the protocol and publication plan. Medtronic reviews publications to determine if confidential information ("CI") is included. Any such CI is deleted before publication. Medtronic may not censor/interfere with the publication. Investigators may publish single-site publications after a decision by Medtronic that no multi-site study publication will be done or 12 months after the study is closed, whichever is earlier.